CLINICAL TRIAL: NCT01872182
Title: A Randomized, Double-Blind, Placebo Controlled, Multicenter, 12-week Phase 3 Study to Evaluate Efficacy and Safety of ALS-L1023 Tablet in Patients With Abdominal Obesity of Metabolic Syndrome
Brief Title: Efficacy and Safety Study of ALS-L1023 in Patients With Abdominal Obesity of Metabolic Syndrome
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-MELS-301
Record Dates: First submitted 2013-05-30; First posted 2013-06-07 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Abdominal Obesity Metabolic Syndrome
MeSH Terms: conditions — Abdominal obesity metabolic syndrome | interventions — ALS-L1023

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test arm (Experimental): ALS-L1023 300mg in two tablets
  Interventions: Drug: ALS-L1023
- Comparator arm (Placebo Comparator): placebo in two tablets
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ALS-L1023 — daily twice for 12 weeks
  Arms: Test arm
Drug: placebo — daily twice for 12 weeks
  Arms: Comparator arm

SUMMARY:
The main objective of this study is to evaluate efficacy and safety of ALS-L1023 tablet in patients with abdominal obesity of metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20 and 64 years(Both genders)
* more than 2 among components of the metabolic syndrome

  * Triglyceride >= 150mg/dL
  * HDL-D: Women < 50mg/dL or Men < 40mg/dL
  * Hypertension: Systolic blood pressure >= 130mmHg or Diastolic blood pressure >= 85mmHg
  * Hyperglycemia: fasting plasma glucose >= 100 mg/dL
* Informed consent awarding

Exclusion Criteria:

* Alcohol or any drug abuse
* Any investigational medication during the preceding 3 months

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2013-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline to 12 week in visceral fat area measured by CT | baseline and 12 week

SECONDARY OUTCOMES:
improvement of metabolic profile | baseline and 12 week
change of insulin resistance | baseline and 12 week
change of BMI | baseline and 12 week

CONTACTS AND LOCATIONS:
Overall Officials: Hye Soon Park, M.D., Ph.D., M.P.H., Principal Investigator — Asan Medical Center
Locations (1):
- 5 Institutions, Seoul, South Korea